CLINICAL TRIAL: NCT04476212
Title: Prophylaxis of Surgical Wound Infection With Topical Antibiotics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Granollers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 20171013
Record Dates: First submitted 2019-01-31; First posted 2020-07-20 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Surgical Site Infection; Surgery--Complications; Colorectal Surgery; Cesarean Section; Infection; Hernia, Abdominal
Keywords: Surgical site infection; Prevention; Topical prophylaxis; Wound irrigation; Topical antibiotic prophylaxis; Abdominal surgery
MeSH Terms: conditions — Surgical Wound Infection; Infections; Hernia, Abdominal | interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Intervention Model Description: It is a randomized, controlled, multicenter, blind study by observer and patient, with two parallel study groups, phase IV. The irrigation of the wound with 0.9% physiological serum will be compared with the irrigation with a solution of amoxicillin-clavulanate, administered topically and dissolved in saline.
Who Masked: Participant, Care Provider, Investigator
Masking Description: There will be masking for the patient, for the surgeon responsible for the case, for the investigator responsible for each study, for the coordinator of the center and for the main investigator. After the closure of the abdominal fascia, the patients will be randomized to one of the study groups. The circulating nurse will open the randomization envelope and prepare the solution indicated on the outside of the operating room. He/she will record the case on the database and will be the only person with knowledge of the group allocation of the case.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In the experimental arm, the surgical wound will be irrigated using an antibiotic solution (amoxicillin-clavulanate) for topical prophylaxis
  Interventions: Other: Topical antibiotic prophylaxis
- Control (No Intervention): In the control arm, the surgical wound will be irrigated with saline, which is our routine at present.

INTERVENTIONS:
Other: Topical antibiotic prophylaxis — The surgical wound will be irrigated with an antibiotic solution, and then we will apply the same solution using gauze for two minutes on the wound
  Arms: Intervention

SUMMARY:
Surgical site infection (SSI) is the main complication of surgery. The prevention of superficial SSI by topical prophylaxis is controversial. Human studies on wound lavage with topical solutions (saline, antiseptics or antibiotics) are old and do not yield conclusive results. In experimental conditions there is evidence in favor of the efficiency wound lavage with saline and antibiotic solutions. Clinical studies are needed to demonstrate the safety and efficacy of antibiotic lavage. Objective. Study of the efficacy of topical antibiotic therapy in the prevention of SSI in patients undergoing abdominal surgery with different risk of infection. Method. Project comprising several randomized double-blind clinical trials with a common methodology. Procedures with varying degrees of contamination, as emergency abdominal surgery, cesareans and complex abdominal wall reconstructions will be studied. Follow-up will be 30 days after operation. Data will be collected anonymously and the relationships between the variables will be analyzed using Pearson's chi-square, survival analysis and analysis of risk factors as appropriate. The effect of topical antibiotic on hospital stay, resistance patterns in SSI, and antibiotic serum levels will be analyzed.

DETAILED DESCRIPTION:
Several Surgical site infection (SSI) prevention guidelines have been published over the last 10 years. Topical prophylaxis of the surgical wound with antibiotics or antiseptics is one of the most controversial measures proposed for SSI prevention. Two guidelines (British, Spanish Ministry of Health) explicitly recommend not irrigating surgical wounds with any product. The World Health Organization considers irrigation with antibiotics as an unresolved issue and, together with the Centers for Disease Control, recommends irrigation with a solution of povidone iodine. The other four guides do not mention the measure. In Catalonia, a SSI prevention bundle recommends wound irrigation with saline, with a low level of recommendation.

Therefore, topical prophylaxis with operational wound washings with different solutions has been poorly studied, evokes contradictory recommendations and is not included in the majority of clinical practice guidelines for SSI prevention.

However, there we detected a high level of use of wound irrigation at the end of an intervention in actual clinical practice. In a survey conducted by 2017 by our group and answered by 845 general surgeons of the Spanish Association of Surgeons, before closing the skin, most surgeons (80.6%) irrigate the subcutaneous layer of the wound, either with saline (51.2%), an antiseptic solution (23.8%) or an antibiotic solution (1.5%). Only 19.4% of respondents do not irrigate. In another survey in 2018, focused on colorectal surgeons of two Spanish associations, similar rates of irrigation with saline, antiseptic or antibiotic were used (55%, 28.9% and 2.2%, respectively) The hypothesis of the study is that topical prophylaxis of the surgical wound with irrigation with an antibiotic solution decreases the rate of postoperative infection in patients undergoing abdominal surgery with different levels of contamination.

The study will compare the efficacy of topical prophylaxis in the surgical wound with an irrigation with an antibiotic solution in the incidence of SSI in abdominal surgery.

It is a randomized, controlled, multicenter, blind study by observer and patient, with two parallel study groups, phase IV.

Design of studies The project includes several prospective comparative studies on the effect of irrigation of surgical wounds with an antibiotic solution on the incisional SSI rate in abdominal surgery. The studies share a unique methodology applied to various types of abdominal surgery with different expected SSI rates and different risk factors.

In the trials, the irrigation of the wound with 0.9% physiological serum will be compared with the irrigation with an active principle solution of a pharmaceutical specialty of proven efficacy by parenteral route, administered topically and dissolved in physiological serum.

Four studies on different types of operations are defined according to the risk of infection:

* Study 1. Complex abdominal wall surgery
* Study 2. Cesarean section
* Study 3. Colorectal elective surgery
* Study 4. Emergency abdominal surgery For each study two groups will be formed, the study group (irrigation with antibiotic solution) and the control group (irrigation with saline).

The project has received the Spanish Drug Agency authorization as a low intervention study, a grant from the Spanish Ministry of Health and the Ethics Committee authorization of the Hospital General of Granollers.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for elective abdominal wall surgery by open route
* Patients admitted for urgent or elective cesarean section
* Patients undergoing elective surgery of the colon or rectum for neoplastic pathology (open or laparoscopy)
* Patients undergoing emergency abdominal surgery (open or laparoscopy)

Exclusion Criteria:

* Patients under treatment with immunosuppressors, corticosteroids and patients on hemodialysis
* Patients with primary peritonitis and liver cirrhosis
* Patients with suspected allergy to the antibiotic used in the study
* Patients who have recently undergone open abdomen surgery (up to 30 days pre-intervention) or to which the wound can not be closed surgical according to the surgeon's criteria
* Patients with American Society of Anaesthesiology classification 5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2018-12-27 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Site infection rate | 30 days
  signs of infection at any level of surgical site

SECONDARY OUTCOMES:
Complications after surgery | 30 days
  Any complication after surgery, evaluated by the Clavien-dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Josep Maria Badia, PhD, Principal Investigator — Fundació Privada Hospital Asil de Granollers; Felipe Ojeda, PhD, Principal Investigator — Fundació Privada Hospital Asil de Granollers
Locations (1):
- Fundació Privada Hospital Asil de Granollers, Granollers, Barcelona, Spain